CLINICAL TRIAL: NCT02994797
Title: Elastometry of the Salivary Glands in Sicca Syndrome
Brief Title: Ultrasound Elastography of Salivary Glands
Acronym: ELSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ELSA
Record Dates: First submitted 2016-07-07; First posted 2016-12-16 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2018-08

CONDITIONS: sjögren Disease
Keywords: salivary glands; ultrasonography; elastometry; elastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ultrasonography in salivary gland has demonstrated its usefulness to diagnose and follow patients with Sjögren syndrome (pSS). More recently, a new imaging technique allows to study the parenchymal elasticity in salivary glands and could be a new tool to evaluate patients with sicca syndrome and pSS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* More than 18 years old
* Consulting in Doppler unit for sicca syndrome or suspicion of Sjögren syndrome
* Consent agreement

Exclusion Criteria:

* No consent agreement
* No sicca symptoms

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female
  more than 18 years old
  consulting in Doppler unit for sicca syndrome or suspicion of Sjögren syndrome
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
salivary glands elastometry | 1 day
  Measure of elasticity of salivary glands (parotid, submandibular and sublingual) in centimeter per second

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No